CLINICAL TRIAL: NCT00668850
Title: A 26-Week, Open-Label, Randomized, Active Comparator Study of Generex Oral-lyn™ Spray and Injected Human Insulin In Subjects With Type-1 Diabetes Mellitus
Brief Title: Active Comparator Study of Generex Oral-lyn™ Spray and Injected Human Insulin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Generex Biotechnology Corp. (Industry)
Collaborators: OSMOS Clinical Research, Inc (Other); PSI Pharma Support Intl (Unknown); Nextrials, Inc. (Industry); eResearch Technology, Inc. (Industry); Hoffmann-La Roche (Industry); ACM Pivotal Global Central Laboratory (Industry)
Responsible Party: George E. Markus, Generex Biotechnology Corp.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN-084-OL
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Generex Oral-lyn™ spray in a split-dose fashion (half the dose immediately prior to the meal and half the dose immediately after the meal) + BID NPH insulin AM and PM as pre-randomization dose
  Interventions: Drug: Generex Oral-lyn™
- 2 (Active Comparator): Regular human insulin 30 minutes before meals + BID NPH insulin AM and PM as pre-randomization dose.
  Interventions: Drug: Regular human insulin

INTERVENTIONS:
Drug: Generex Oral-lyn™ — Generex Oral-lyn™ spray in a split-dose fashion (half the dose immediately prior to the meal and half the dose immediately after the meal) + BID NPH insulin AM and PM as pre-randomization dose
  Other Names: buccal Insulin spray
  Arms: 1
Drug: Regular human insulin — Regular human insulin 30 minutes before meals + BID NPH insulin AM and PM as pre-randomization dose.
  Other Names: insulin
  Arms: 2

SUMMARY:
To compare the efficacy of Generex Oral-lyn™ RapidMist™ System and standard regular human insulin therapy as measured by HbA1c, in type-1 diabetes mellitus subjects on BID NPH intermediate acting insulin therapy.

DETAILED DESCRIPTION:
This is a 26 week open-label, randomized, multi-center, active comparator study to compare oral spray insulin (Generex Oral-lyn™) with regular human insulin therapy as measured by HbA1c, and number of hypoglycaemic episodes in type-1 diabetes mellitus subject. All subjects will be on BID NPH intermediate acting insulin therapy. If subject is using long acting insulin (Glargine, Detemir, etc.), he/she must be switched to NPH intermediate acting insulin. If on insulin analogue (Novolog, Lispro, Aspart, Aphidra, Glulisine, or any other analogue available in the subject's geographical area), the subject must be switched to regular human insulin 3 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female between the ages 18 to 75 years
* Type 1 diabetes mellitus patients (according to ADA and/or WHO classification) who have >1 year history of type 1 DM and are currently managed with daily insulin injections totalling 0.3 to 0.8 IU/kg of body weight;
* Current physical examination, vital signs and ECG at screening that reveals no clinically significant abnormalities;
* Have a body mass index (BMI) <27;
* 8.5% (inclusively)<Have a glycosylated haemoglobulin HbA1c
* Willing and able to follow the American Diabetes Association diet guidelines for type 1 diabetes; be able to commit to perform home blood glucose monitoring and record values as well as hypoglycemic events
* Willing to give written informed consent prior to admission into the study.

Exclusion Criteria:

* Have a significant active asthma or suspected abnormalities of buccal mucosa; cardiovascular, cerebrovascular, hepatic, renal, gastrointestinal, hematological, or auto-immune disease (other than auto-immune thyroid disease); history of athopy or drugs allergy
* Have evidence of unstable retinopathy (defined as pre-proliferative or proliferative retinopathy currently requiring photocoagulation therapy), nephropathy or neuropathy (gastroparesis or orthostatic hypotension);
* Have hypoglycemia unawareness;
* Have had more than one episode of severe hypoglycemia with seizure or coma or ketoacidosis within the past 12 months;
* Have a blood pressure in excess of 160/100 mmHg at the Screening visit;
* Have had any acute illness within the 2 weeks prior to screening;
* Have a history of drug or alcohol abuse that in the opinion of the Investigator would interfere with participation in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of Generex Oral-lyn™ RapidMist™ System and standard regular human insulin therapy as measured by HbA1c, in type-1 diabetes mellitus subjects on BID NPH intermediate acting insulin therapy | change in HbA1c from the Day 0 (V3) to Day 180 (V9) of Treatment Phase.

SECONDARY OUTCOMES:
To evaluate the safety, tolerability, and satisfaction with Generex Oral-lyn™ therapy when administered by the RapidMist™ Diabetes Management System | 26 week

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Bernstein,, MD, Study Chair — Generex Biotechnology Corp.; Jaime Davidson, MD, Study Director — Generex Biotechnology Corp.; Philip Raskin, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (74):
- United States (8):
  - Coastal Biomedical Research Inc. at Santa Monica, 2001 Santa Monica Blvd Suite 390W, California
  - The Center for Diabetes & Endocrine Care at Hollywood, 1150 N. 35th Ave Suite 590, Florida
  - Physicians Research Group at Indianapolis, 7400 North Shadeland Ave, Indiana
  - MODEL Clinical Research at Baltimore, 6535 North Charles Street Suite 400N, Maryland
  - Grunberger Diabetes Institute at Bloomfield Hills, 43494 Woodward Ave Suite 208, Michigan
  - Beth Israel Medical Center, Geral J. Friedman Diabetes Institute at New York, 317 East 17th Street Room 7F05 8th Floor, New York
  - Multiple Health Research, LLC. at Arlington, 501 Rita Lane Suite 113, Texas
  - University of Texas Southwestern Medical Center at Dallas, 5323 Harry Hines Blvd, Texas
- Bulgaria (6):
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska", 1 Saint Georgi Sofiysky Saint, Sofia
  - University Multiprofile Hospital for Active Treatment at Varna, 1 Hristo Smirnensky Saint
  - Multiprofile Hospital for Active Treatment at Stara Zagora, 11 Armeyska Saint
  - University Multiprofile Hospital for Active Treatment at Plovdiv, 15A Vassil Aprilov Blvd
  - Multiprofile Hospital for Active Treatment at Ruse, 2 Nezavisimost Saint
  - University Multiprofile Hospital for Active Treatment at Pleven, 8A Georgi Kotchev Saint
- Canada (3):
  - The Bailey Clinic at Red Deer, #108 3947 50A Avenue, Alberta
  - Calgary Metabolic Education & Research Centre at Calgary, #23, 4411-16th Avenue Northwest, Alberta
  - West Edmonton Diabetes Centre, 10230 142 Saint Northwest # 25, Edmonton, Alberta
- Instituto de Endocrinologia IEMYR, Avenida La Coruña Nº 6337 Y San Ignacio, Quito, Ecuador
- Poland (9):
  - Bydgoszcz Diabetology and Endocrinology Center at Bydgoszcz, Ul. Baczynskiego 17
  - OSTEOMED Medical Center at Warszawa, Ul. Bialobrzeska 40A
  - Chair and Department of Internal Medicine and Diabetology, Voivodship Brodnowski Hospital at Warszawa, Ul. Kondratowicza 8
  - Diabetology Clinic for Adults, NZOZ Elblag Diabetology Center, Ul. Krolewiecka 146
  - TeMeD - Clinical Trials at Rzeszow, Ul. Mazowiecka 56
  - Provincial Centre of Diabetology and Metabolic Diseases, M.Pirogow Provincial Specialist Hospital at Lodz, Ul. Nowa 30/32
  - Silesia Osteoporosis Center at Katowice, Ul. Opolska 11/3
  - TeMeD - Clinical Trials at Nowy Targ, Ul. Wojska Polskiego 14
  - NZOZ Specialist Centre of Internal Medicine and Diabetology Malgorzata Arciszewska at Bialystok, Ul. Zamenhofa 10/20
- Puerto Rico (3):
  - Celis Aguilera 10B, Fajardo
  - Puerto Medical Center, San Juan
  - Clinical Research, Puerto Rico, San Juan
- Romania (9):
  - "Nicolae Malaxa" Clinical Hospital, Department of Diabetes, Nutrition and Metabolic Diseases at Bucharest, 12 Vergului Saint Sector 2
  - Timisoara Emergency Clinical County Hospital, Clinic of Diabetes, Nutrition and Metabolic Diseases at Timisoara, 156 Iosif Bulbuca Av
  - Satu Mare County Hospital, Department of Diabetology and Nutrition Diseases at Satu Mare, 2-3 Eroii Revolutiei Square
  - Private Practice at Galati, 25 Constructorilor St, Bl. E5/64
  - Cluj Emergency Clinical County Hospital, Department of Diabetes, Nutrition and Metabolic Diseases at Cluj-Napoca, 3-5 Clinicilor Saint
  - Oradea Clinical County Hospital, Department of Diabetes, Nutrition and Metabolic Diseases at Oradea, 33 Republicii Saint
  - National Institute of Diabetes, Nutrition and Metabolic Diseases, 1st Clinical Department of Diabetes, Nutrition and Metabolic Diseases at Bucharest, 5-7 Ion Movila Saint Sector 2
  - Cardiology Private Practice at Bala Mare, 6/72 Independentei Saint
  - Private Practice Nicodiab SRL at Bucharest, 92 Polona St, Bl 17 A+B, Sc. 1, Ap. 2
- Russia (27):
  - Municipal Medical Institution: City Hospital # 2, Municipal Diabetology and Rehabilitation Center, 1 3rd -Transportnaya Str., Omsk
  - St. Petersburg State Medical Institution: St. George Municipal Hospital, 1 Severny Pr., St.Petersburg
  - Municipal Medical Institution: Medical Unit "Izhmash", Municipal Endocrinology Center, 1 Truda Str., Izhevsk
  - St. Petersburg State Medical Institution: Municipal Consulting and Diagnostic Center #1, St. Petersburg Territorial Diabetology Center, 10 Siqueirosa Str., Saint Petersburg
  - Federal State Institution: Endocrinology Research Center under the Federal Agency for High-Tech Medical Care, Department of Therapeutic and Surgical Methods for Treatment of Diabetic Foot, 11 Dmitriya Ulyanova Str., Moscow
  - Federal State Institution: Endocrinology Research Center under the Federal Agency for High-Tech Medical Care, Department of Training and Psychosocial Rehabilitation of Patients with Diabetes Mellitus, 11 Dmitriya Ulyanova Str., Moscow
  - St. Petersburg State Medical Institution: Municipal Hospital of St. Elizabeth, 14 Vavilovykh Str., Saint Petersburg
  - State Medical Institution: Nizhny Novgorod Regional Clinical Hospital n.a. N.A. Semashko, 190 Rodionova Str., Nizhny Novgorod
  - Medical Institution Municipal Clinical Hospital #67, 2 "b" Salyama Adilya Str., Moscow
  - State Medical Institution: Kemerovo Regional Clinical Hospital, 22 Oktyabrsky Pr., Kemerovo
  - State Medical Institution: Arkhangelsk Regional Clinical Hospital, 292 Lomonosova Pr., Arkhangelsk
  - State Medical Institution: Republican Hospital, 3 Pirogova Str., Petrozavodsk, ,
  - St. Petersburg State Medical Institution:Municipal Outpatient Clinic #51, 33/35 Kosmonavtov Pr., Saint Petersburg
  - Moscow State Medical Institution Municipal Clinical Hospital #68, 4 Shkuleva Str., Moscow
  - St. Petersburg State Medical Institution: City Aleksandrovskaya Hospital, 4 Solidarnosti Pr., Saint Petersburg
  - Federal State Medical Institution: All-Russia Center for Urgent Care and Radiation Medicine n.a. A.M. Nikiforov under the Russian Emergency Control Ministry, 4/2 Lebedeva Str., St.Petersburg
  - St. Petersburg State Medical Institution: Municipal Multifield Hospital #2, 5 Uchebny Per., Saint Petersburg
  - State Higher Educational Institution: Tyumen State Medical Academy under the Federal Agency for Healthcare and Social Development, Multifield Clinic, 54 Odesskaya Str., Tyumen
  - "Diabetes" Center Company Limited, 56 Sovetskoi Armii Str., Samara
  - State Medical Institution: Consulting and Diagnostic Center of Komi Republic, Diabetology Center, 6 Kuratova Str., 167981
  - State Medical Institution: Murmansk Regional Consulting and Diagnostic Center, 6 Pavlova Str., Building 4, Murmansk
  - Municipal Medical Institution: Municipal Clinical Hospital #1, Municipal Diabetology Center, 6 Zalesskogo Str., Novosibirsk
  - State Higher Educational Institution: St. Petersburg State Medical University n.a. I.P. Pavlov under the Federal Agency for Healthcare and Social Development, 6/8 L. Tolstogo Str., Saint Petersburg
  - State Institution: Moscow Regional Research Clinical Institute n.a. M.F.Vladimirsky, 61/2 Shchepkina Str., Moscow
  - State Higher Educational Institution: Ural State Medical Academy under the Federal Agency for Healthcare and Social Development; Family Medicine Clinic, 7 Kluchevskaya Str., Ekaterinburg
  - State Medical Healthcare Institution: Chelyabinsk Regional Clinical Hospital, 70 Vorovskogo Str., Medgorodok, Chelyabinsk
  - State Medical Institution:Territorial Endocrinology Center, Territorial Diabetology Center, 9 Artema Str., Stavropol
- Ukraine (8):
  - Regional Endocrinology Center, Diabetology Department at Lviv, 1, Ostrozskoho St., Lviv
  - Ukrainian Research and Development Center for Endocrine Surgery and Endocrine Organ and Tissue Transplantation under the Ministry of Health of Ukraine, General Endocrine Pathology Department at Kiev, 121, Kharkovskoe Shosse, Kiev
  - M.V. Sklifosovskyi Regional Clinical Hospital, Endocrinology Department at Poltava, 23, Shevchenko Saint
  - City Clinical Hospital #9, Endocrinology Department at Dnipropetrovsk, 29, Vorontsova Saint
  - M.O. Semashko Republican Clinical Hospital, Endocrinology Department at Simferopol, 69 Kievskaya Saint
  - V.P. Komisarenko Institute for Endocrinology and Metabolism under the Ukrainian Academy of Medical Sciences, Clinical Diabetology Department at Kiev, 69, Vyshgorodskaya St., Kiev
  - V.P. Komisarenko Institute for Endocrinology and Metabolism under the Ukrainian Academy of Medical Sciences, General Endocrine Pathology Department at Kiev, 69, Vyshgorodskaya St., Kiev
  - V.Ya. Danylevskyi Institute for Endocrine Pathology under the Ukrainian Academy of Medical Sciences, Clinical Endocrinology Department at Kharkov, Pomerky 27, Kharkov